CLINICAL TRIAL: NCT00567450
Title: Ropivacaine 0.75% vs Ropivacaine 0.75% Plus Mepivacaine 1.5% for Subgluteal Sciatic Bloc: a Prospective Double Blind Randomized Controlled Study
Brief Title: Ropivacaine Versus Ropivacaine Plus Mepivacaine for Sciatic Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Prof Herve Dupont, Anesthesiology and Critical Care Department
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2007-002254-31; EudraCT: 2007-002254-31; AFFSAPS: A70388-33
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Subgluteal Sciatic Block
Keywords: sciatic block; ropivacaine; mepivacaine; locoregional anesthesia
MeSH Terms: interventions — Ropivacaine; Mepivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- B (Active Comparator): 30ml of a mixture of ropivacaïne 0.75% associated with mepivacaïne 1.5%
  Interventions: Drug: ropivacaine plus mepivacaine
- A (Experimental): 30 ml of ropivacaine 0.75%
  Interventions: Drug: ropivacaine

INTERVENTIONS:
Drug: ropivacaine — 30ml of a mixture of ropivacaïne 0.75%
  Arms: A
Drug: ropivacaine plus mepivacaine — 30ml of a mixture of ropivacaïne 0.75% associated with mepivacaïne 1.5%
  Arms: B

SUMMARY:
In loco regional anesthesia, much more than for general anesthesia, the choice of the product is largely left at the discretion of the practitioner. Two categories of local anesthetics are distinguished according to their pharmacodynamic characteristics: products with a short time of installation and a short duration period, and products with a longer delay of installation of the sensitive and motor block, but with a long-term duration. Indeed, the combined use of two products pharmacodynamically different seems to be of a practical interest.

This study provides a comparison of the onset of action of 30 ml of ropivacaine 0.75% and 30ml of a mixture of ropivacaïne 0.75% associated with mepivacaïne 1.5% for the subgluteal sciatic nerve block. This is a prospective randomized double-blind study where the main criterion of judgment is the time of installation of a sensitive block compatible with surgery in the sciatic territory nerve. Fifteen patients per group were calculated to detect a 50% decrease of the onset of action in the combination group with a power of 90% and alpha to 5%, according to a previous pilot study. The secondary endpoints are the intensity and time of installation of the motor block, the duration of sensitive and motor block, the total dose of morphine administered within 48 hours, as well as its possible side effects.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* surgery of the foot under sciatic block

Exclusion Criteria:

* no indication of locoregional anesthesia
* polyneuropathy or any neurological disease
* know hypersensitivity to local anesthetics
* porphyria
* atrio-ventricular block
* not controlled epilepsia
* hypovolemia
* pregnancy
* anticoagulant treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Time of installation of a sensitive block compatible with surgery in the sciatic territory nerve | 4h

SECONDARY OUTCOMES:
intensity and time of installation of the motor block, the duration of sensitive and motor block, the total dose of morphine administered within 48 hours, and its side effects. | 48h

CONTACTS AND LOCATIONS:
Overall Officials: Campana Philippe, MD, Principal Investigator — Anesthesiology department
Locations (1):
- CHU d'Amiens, Pole Anesthesie Réanimation, Place Victor Pauchet, Amiens, France